CLINICAL TRIAL: NCT05266027
Title: The Efficacy of Long-Acting Nalbuphine Sebacate (Naldebain) for Pain Management After Knee Arthroplasty
Brief Title: Naldebain for Pain Management After Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20210150
Record Dates: First submitted 2022-02-20; First posted 2022-03-04 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2022-11

CONDITIONS: Arthropathy of Knee Joint

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Nalbuphine Sebacate (Naldebain) intramuscular injection
  Interventions: Drug: Nalbuphine Sebacate (Naldebain)
- Placebo Group (Placebo Comparator): Placebo medication intramuscular injection
  Interventions: Drug: Placebo medication

INTERVENTIONS:
Drug: Nalbuphine Sebacate (Naldebain) — Nalbuphine Sebacate (Naldebain) 2mL/150mg would be intramuscularly injected during knee arthroplasty surgery.
  Arms: Experimental Group
Drug: Placebo medication — Placebo medication, Nalbuphine Sebacate not contained
  Arms: Placebo Group

SUMMARY:
Naldebain, a long-acting analgesic injection, obtained a license from the Taiwan Food and Drug Administration (TFDA) of the Ministry of Health and Welfare on March 6, 2017 to approve a sustained-release long-acting analgesic on the market in Taiwan. This study hopes to use a rigorous double-blind randomized controlled experiment to understand whether the new sustained-release analgesic Naldebain can achieve effective pain relief for patients undergoing knee replacement surgery, and to evaluate the patient's functional recovery status .

DETAILED DESCRIPTION:
Naldebain, a long-acting analgesic injection, obtained a license from the Taiwan Food and Drug Administration (TFDA) of the Ministry of Health and Welfare on March 6, 2017 to approve a sustained-release long-acting analgesic on the market in Taiwan. At present, it is the only analgesic injection that has an efficacy of up to seven days. The currently approved drug indication is to relieve moderate and severe acute pain after surgery. Pharmacological mechanisms and experiments show that its analgesic effect is equivalent to morphine, but its side effects are much lower than morphine. Because of its special pharmacological mechanism, it has extremely high potential to improve patients undergoing knee replacement surgery. Therefore, this study hopes to use a rigorous double-blind randomized controlled experiment to understand whether the new sustained-release analgesic Naldebain can achieve effective pain relief for patients undergoing knee replacement surgery, and to evaluate the patient's functional recovery status .

ELIGIBILITY:
Inclusion Criteria:

* Age at least 50 years old, not exceed 100 years old
* Diagnosed Primary Knee Osteoarthritis accepted Knee Arthroplasty

Exclusion Criteria:

* Diagnosed inflammatory Arthritis、Rheumatoid Arthritis
* Accepted Revision Knee Arthroplasty
* Patients with head injury, intracranial injury, increased intracerebral pressure and liver insufficiency
* Patients who are allergic to nalbuphine sebacate, nalbuphine, sesame oil or benzyl benzoate drugs

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
The amount of painkillers used by the Patient Controlled Analgesia machine (PCA machine) | Post operation Day1
  morphine consumption amount
The amount of painkillers used by the Patient Controlled Analgesia machine (PCA machine) | Post operation Day2
  morphine consumption amount
The amount of painkillers used by the Patient Controlled Analgesia machine (PCA machine) | Post operation Day3
  morphine consumption amount
The level of pain index (Visual Analog Scale) | Baseline
  pain level, Visual Analog Scale higher scores mean a worse outcome, 0~10
The level of pain index (Visual Analog Scale) | Post operation Day1
  pain level, Visual Analog Scale higher scores mean a worse outcome, 0~10
The level of pain index (Visual Analog Scale) | Post operation Day2
  pain level, Visual Analog Scale higher scores mean a worse outcome, 0~10
The level of pain index (Visual Analog Scale) | Post operation Day3
  pain level, Visual Analog Scale higher scores mean a worse outcome, 0~10
The level of pain index (Visual Analog Scale) | Post operation Day4
  pain level, Visual Analog Scale higher scores mean a worse outcome, 0~10
The level of pain index (Visual Analog Scale) | Post operation Day5
  pain level, Visual Analog Scale higher scores mean a worse outcome, 0~10
The level of pain index (Visual Analog Scale) | Post operation 2 weeks
  pain level, Visual Analog Scale higher scores mean a worse outcome, 0~10
The level of pain index (Visual Analog Scale) | Post operation 6 weeks
  pain level, Visual Analog Scale higher scores mean a worse outcome, 0~10

SECONDARY OUTCOMES:
knee joint functional data questionnaire (Western Ontario and McMaster Universities Osteoarthritis Index) | Baseline
  knee joint functional data questionnaire
knee joint functional data questionnaire (Western Ontario and McMaster Universities Osteoarthritis Index) | Post operation 2 weeks
  knee joint functional data questionnaire
knee joint functional data questionnaire (Western Ontario and McMaster Universities Osteoarthritis Index) | Post operation 6 weeks
  knee joint functional data questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hsuan-Ti Huang, M.D., Study Director — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No